CLINICAL TRIAL: NCT04522375
Title: A Multinational, Multicenter, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Activity of FP 045 in Patients With Fanconi Anemia (FusuciA Study)
Brief Title: A Dose Escalation Study of FP-045 in Patients With Fanconi Anemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Twenty months after investigative site initiations, and best efforts to identify study participants, no participants were identified.
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP045C-19-001
Record Dates: First submitted 2020-08-03; First posted 2020-08-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Intervention Model Description: Phase of dose escalation to OBD followed by 3 months of treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FP-045 (Experimental): The study will enroll a total of 6 young adult/adolescent patients progressing through three dose levels, followed by a minimum of 8 and up to 12 pediatric patients progressing through up to three dose levels.
  Interventions: Drug: FP-045

INTERVENTIONS:
Drug: FP-045 — activator of aldehyde dehydrogenase

SUMMARY:
This is a multi-center, Phase 1/2 study to determine the Optimal Biologic Dose (OBD) and to evaluate the safety, tolerability, PK, and preliminary activity of FP 045 when administered orally in young adult/adolescent and pediatric patients with Fanconi anemia. The study will enroll a total of 4 young adult/adolescent patients and a minimum of 8 and up to 12 pediatric patients with mild-moderate bone marrow failure who have not undergone hematopoietic cell transplant. This makes the total patient number between 12-16 total. Dose escalation will occur individually for each patient, within each age group. Each patient will receive each of 3 dose levels of FP 045 (intra-patient dose escalation), beginning with Dose Level 1, followed by Dose Levels 2 and 3. Each dose level will be administered for 28 days prior to escalation to the next higher dose level for that patient.

DETAILED DESCRIPTION:
Dose escalation will begin with young adult/adolescent patients. The initial two patients enrolled in the study will be > 15 years of age. These patients must complete the entire 28-day period of treatment at Dose Level 1 prior to additional young adult/adolescent patients being enrolled. All 4 young adult/adolescent patients must complete 28 days of treatment at Dose Level 1, and cumulative safety must be reviewed by the Safety Review Committee (SRC), prior to the enrollment of pediatric patients. The initial two pediatric patients enrolled will be > 6 years of age. These patients must complete the entire 28-day period of treatment at Dose Level 1 prior to additional pediatric patients being enrolled. A minimum of 8 and maximum of 12 pediatric patients will be enrolled to allow for at least 4 patients between the ages of 3-6.

Study assessments will be conducted at each visit. Patients will be observed closely for Dose Limiting Toxicity (DLT) during each dosing period. Any patient experiencing a DLT will have study drug interrupted and will not be allowed to escalate to the next higher dose level. The patient may resume treatment at one dose level lower once the DLT has resolved to baseline or to ≤ Grade 1 in severity. The MTD will be defined as the dose level immediately below the dose level at which DLT occurred. Patients requiring an interruption in treatment of > 3 weeks following a DLT will be withdrawn from the study. The MTD will be assessed separately for each individual patient.

Following the completion of dose escalation, each patient will continue treatment at either the highest dose or their individual MTD, and then transition to the OBD for their age group (once defined), for a total of 3 months. Patients failing to receive 75% of planned doses for reasons other than adverse effects may be replaced.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 3-35
* documented Fanconi anemia by chromosome breakage analysis
* females of child-bearing potential and males required to use highly effective birth control
* mild to moderate bone marrow failure with at least one cytopenia of > grade 1 severity

Exclusion Criteria:

* history of any malignancy except focal squamous cell or basal cell carcinoma of the skin or carcinoma in situ of cervix
* has myelodysplastic syndrome or acute leukemia per world health organization (WHO) criteria
* has history of any significant medical conditions
* has aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 5x upper limit of normal (ULN) or calculated creatinine clearance (Clcr) of < 50 mL/min
* has active Hepatitis B or C
* has an ongoing systemic infection
* requires a strong CYP3A4 inhibitor
* has had major surgery within 30 days
* Active graft versus host disease requiring systemic treatment
* Has a history of bone marrow or stem cell transplant

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Optimal Biologic Dose (OBP) of FP-045 | 28 days x up to 3 doses
  The OBP of FP-045 in adolescent and pediatric subjects
stabilizing or improving cytopenia in FA | 3 months
  Change from baseline in hemoglobin

SECONDARY OUTCOMES:
Safety and tolerability | 3-6 months
  Frequency of adverse events and serious adverse events
pharmacokinetic profile | 3- 6 months
  Mean AUC of FP-045 by dose level

CONTACTS AND LOCATIONS:
Overall Officials: Susan Whitaker, Study Director — Foresee Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — http://clinicaltrials.gov — clinicaltrials.gov
- Available data/document: Statistical Analysis Plan — http://clinicaltrials.gov — clinicaltrials.gov